CLINICAL TRIAL: NCT05813574
Title: Long Term Sequelae of COVID-19: Observational Cohort Study in Twente, the Netherlands
Brief Title: Long Term Impact of COVID-19
Status: Completed | Type: Observational
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: University of Twente (Other); Ziekenhuisgroep Twente (Other)
Responsible Party: Principal Investigator, Harald E. Vonkeman, Principle Investigator, Medisch Spectrum Twente
Other Study IDs: Long COVID
Record Dates: First submitted 2023-04-13; First posted 2023-04-14 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Long COVID-19; Post-COVID-19 Syndrome; COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 survivors: COVID-19 survivors: patients (≥18 years old) who were tested positive for SARS-CoV-2 infection as confirmed by polymerase-chain-reaction (PCR) testing and were subsequently hospitalised, were followed after discharge from hospitals in Enschede (MST), Hengelo or Almelo (ZGT).
  Interventions: Other: Observational patient reported outcomes

INTERVENTIONS:
Other: Observational patient reported outcomes — Of COVID-19 patients

SUMMARY:
COVID-19, caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, has a devastating effect on human lives, including over 6.6 million death as of November 2022. Furthermore, many individuals continue to experience persisting sequelae after the initial infection. Little is known about the impact of undergoing COVID-19 hospitalisation. Hence, the investigators propose an observational longitudinal study in a cohort of COVID-19 survivors after hospital discharge, to examine their perspectives on their health, health-related quality of life, and persistence of common COVID-19 symptoms, such as fatigue, dyspnoea and anxiety. Potential influencing socio-demographic and biological factors will additionally assessed.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥18 years
* PCR-confirmed SARS-CoV-2 infection and hospital admission
* Proficiency in Dutch
* Providing informed consent

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥18 years old) with SARS-CoV-2 infection confirmed by PCR, and hospitalised and subsequently discharged from MST or ZGT hospital
Sampling Method: Non-Probability Sample
Enrollment: 835 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
General health perception | at 12 months after hospital discharge
  measured by Short Form 36 Health Survey (SF-36)

SECONDARY OUTCOMES:
Health-related quality of life | at 3, 6, 9 and 12 months
  measured by Short Form 36 Health Survey (SF-36). Physical role limitations, bodily pain, general health perceptions vitality, social functioning, emotional role limitations and mental health. Min=0, Max=100 where higher scores indicate better health outcomes
Health Status | at 3, 6, 9 and 12 months
  measured by EuroQol 5d(EQ-5D). Mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Min = 1, Max = 5, where higher scores indicate worse health outcomes.
Health Status Scale | at 3, 6, 9 and 12 months
  Measured by EQ Visual Analogue Scale for self-rated health. Min = 0, Max = 100, where higher scores indicate better health outcomes.
Positive Health | at 3, 6, 9 and 12 months
  measured by my Positive Health]): Min = 0, Max = 10, where higher scores indicate better health outcomes
Incidence, severity and course of Fatique | at 3, 6, 9 and 12 months
  measured by Short Fatique Questionnaire; min = 4, max = 28, higher scores indicating worse fatigue]
Incidence, severity and course of Dyspnoea | at 3, 6, 9 and 12 months
  measured by modified Mental Research Council (mMRC) scale; min = 1, max = 6, higher scores indicating worse dyspnoea
Incidence, severity and course of Sleep | at 3, 6, 9 and 12 months
  measured by unvalidated single-item question min = 1, max = 5, higher scores indicating worse sleep
Incidence, severity and course of Post-Traumatic Stress Disorder | at 3, 6, 9 and 12 months
  measured by PTSD checklist for th DSM-5 (PCL-5) COVID-19 version
Experience sampling study measuring fatigue | Six times a day over 14 days
  Fatigue (physical, and mental), 1-7, as single-item with higher scores indicating worse health outcomes
Experience sampling study measuring dyspnoea | Six times a day over 14 days
  Dyspnoea (1 - 7), as single-item with higher scores indicating worse health outcomes
Experience sampling study measuring cognitive functioning | Six times a day over 14 days
  cognitive functioning, 0 - 10, as single-item with higher scores indicating worse health outcomes
Experience sampling study measuring pain | Six times a day over 14 days
  pain (headache, joint pain, chest pain or discomfort, and pain elsewhere/non-specific; 0 - 10, as single-item with higher scores indicating worse health outcomes
Experience sampling study measuring severity and daily course of positive and negative affect | Six times a day over 14 days
  Positive (excited, relaxed, satisfied, thankful, and happy) and negative (anxious, gloomy, sad, irritable, and disappointed) affect (all single-items; 1 - 7, higher scores indicating better and worse outcomes for positive and negative affect respectively
Experience sampling study measuring daily activity | Six times a day over 14 days
  Type of activity just before measurement; o Options: 1: nothing; 2: strenuous relaxation (for example walking, riding a bike, gardening); 3: passive relaxation (for example watching television, reading a book); 4: sleeping or resting; 5: Work/study; 6: household chores; 7: Eating/drinking; 8: self-care (for example bodily hygiene, medication); 9: On the go; 10: social interaction; 11: Something else, namely…
Experience sampling study measuring sleep | Once a day for 14 days
  Sleep (quality and duration) ; single-item; How many hours of sleep did you get last night?
Experience sampling study measuring naps | Once a day for 14 days
  naps (frequency and duration; single-item
Experience sampling study measuring health status | Once a day for 14 days
  Self-reported health status (EQ-VAS of the EQ-5D-5L; 0 - 100; higher scores indicating better health outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Harald E. Vonkeman, PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Background] Wensink M, Schaap G, Ten Klooster PM, Doggen CJM, van der Palen J, Vonkeman HE, Bode C. Physical and mental fatigue in post-COVID syndrome and their associations over time: A small-sample ESM-study to explore fatigue, quality of sleep and behaviours. J Psychosom Res. 2023 Jan;164:111084. doi: 10.1016/j.jpsychores.2022.111084. Epub 2022 Nov 17. PMID 36436226
- [Background] Schaap G, Wensink M, Doggen CJM, van der Palen J, Vonkeman HE, Bode C. "It Really Is an Elusive Illness"-Post-COVID-19 Illness Perceptions and Recovery Strategies: A Thematic Analysis. Int J Environ Res Public Health. 2022 Oct 11;19(20):13003. doi: 10.3390/ijerph192013003. PMID 36293582